CLINICAL TRIAL: NCT04531319
Title: Evaluation of Immune Cell Subgroups in Covid 19 Patients
Brief Title: Immune Cell Subgroups in Covid 19 Patients
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, Assoc. Prof., Istanbul Training and Research Hospital
Other Study IDs: Covid Cell
Record Dates: First submitted 2020-08-27; First posted 2020-08-28 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Covid19
Keywords: T helper cell; T cytotoxic cell; Monocyte; NK cell
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: Covid 19 (+) patients
  Interventions: Diagnostic Test: Flow cytometric analysis
- Control Group: Healthy volunteers
  Interventions: Diagnostic Test: Flow cytometric analysis

INTERVENTIONS:
Diagnostic Test: Flow cytometric analysis — Flow cytometric analysis of T helper, T cytotoxic cells, NK cells and monocytes

SUMMARY:
COVID-19, spreading rapidly all over the world, causes serious morbidity and mortality. In severe COVID-19 infections, after pulmonary inflammation, cardiovascular organ failure, cytokine storm, hemophagocytosis, septic shock, develops due to uncontrolled hypoxia, and isolated organ failure turns into multi-organ failure. It is noteworthy that it causes lymphopenia in patients. In studies conducted, the effects of Covid-19 on the immune system were evaluated with limited parameters. In addition, no study evaluating the effect of this disease on the immune system has been published in our country.

DETAILED DESCRIPTION:
The causative agent of coronavirus 2019 (COVID-19) disease, which started in Wuhan province of China in December 2019, was severe acute respiratory failure syndrome coronavirus 2 (SARS-CoV-2), which quickly spread all over the world and caused a pandemic. COVID-19 can cause death with symptoms such as fever, cough, muscle pain, shortness of breath, and pneumonia (1). Pulmonary pathology of COVID-19 is diffuse alveolar damage, focal reactive hyperplasia of pneumocytes with patchy inflammatory cells, intravascular thrombosis, monocyte, macrophage and lymphocyte infiltration into pulmonary spaces. Severe infiltration of pulmonary tissue affects alveolar gas exchange. In addition, cardiovascular morbidity, tachyarrhythmia and thromboembolic events are observed in 1/5 of the hospitalized patients with troponin elevation, which is closely related to mortality. In severe COVID-19 infections, after pulmonary inflammation, cardiovascular organ failure, cytokine storm, hemophagocytosis, septic shock, develops due to uncontrolled hypoxia, and isolated organ failure turns into multi-organ failure.

It is noteworthy that it causes lymphopenia in patients. In the studies conducted, the effects of Covid-19 on the immune system and the determination of cell subgroups were performed with limited parameters. No studies have been conducted on PDL-1, one of the immune control points. In addition, no study evaluating the effect of this disease on the immune system with wide parameters has been published in our country.

We aimed to study CD3 (+) lymphocytes, CD4 (+) lymphocytes, CD 8 (+) lymphocytes, CD 3(-)/CD16 (+) NK cell ratio, CD14 (+) lymphocytes, and HLA-DR positivity on CD14 (+) cells at Covid-19 and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Covid 19 PCR (+) results

Exclusion Criteria:

* Cancer Patients
* Patients with known immunodeficiency
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who admitted to the emergency department with the complaint of respiratory failure, lymphopenia in blood tests and Covid 19 (+) in the PCR tests are case group.
  Also healty volunteers who don't have complaint of respiratory failure, lymphopenia in blood tests and Covid 19 (-) in the PCR tests are control group.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
T cell subtype ratios | 1 month
  T helper, NK cell and T cytotoxic cell ratio

SECONDARY OUTCOMES:
Monocyte ratio | 1 month
  CD14 (+) monocyte and HLA-DR (+) cell ratio

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk Oguz Idiz, Assoc. Prof, Principal Investigator — Istanbul Training and Research Hospital
Locations (1):
- Istanbul Training and Reseach Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bi Q, Wu Y, Mei S, Ye C, Zou X, Zhang Z, Liu X, Wei L, Truelove SA, Zhang T, Gao W, Cheng C, Tang X, Wu X, Wu Y, Sun B, Huang S, Sun Y, Zhang J, Ma T, Lessler J, Feng T. Epidemiology and transmission of COVID-19 in 391 cases and 1286 of their close contacts in Shenzhen, China: a retrospective cohort study. Lancet Infect Dis. 2020 Aug;20(8):911-919. doi: 10.1016/S1473-3099(20)30287-5. Epub 2020 Apr 27. PMID 32353347
- [Background] Felsenstein S, Herbert JA, McNamara PS, Hedrich CM. COVID-19: Immunology and treatment options. Clin Immunol. 2020 Jun;215:108448. doi: 10.1016/j.clim.2020.108448. Epub 2020 Apr 27. PMID 32353634
- [Background] Ganji A, Farahani I, Khansarinejad B, Ghazavi A, Mosayebi G. Increased expression of CD8 marker on T-cells in COVID-19 patients. Blood Cells Mol Dis. 2020 Jul;83:102437. doi: 10.1016/j.bcmd.2020.102437. Epub 2020 Apr 13. PMID 32325421